CLINICAL TRIAL: NCT04909372
Title: Impact of Environmental Labelling on Food Choices : a Randomized Controlled Trial in a Virtual Reality Supermarket
Brief Title: Environmental Labelling in a Virtual Supermarket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EIPH0126
Record Dates: First submitted 2021-05-24; First posted 2021-06-01 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Diet, Healthy; Food Selection
Keywords: labelling; food choice
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No labelling (No Intervention): Food products without any label in the virtual supermarket.
- Environmental labelling (Experimental): Food products with an environmental label in the virtual supermarket.
  Interventions: Behavioral: Labelling

INTERVENTIONS:
Behavioral: Labelling — Food products in the virtual supermarket will display an environmental label on their packaging, from A (lowest impact) to E (highest impact). The label categories are based on the Product Environmental Footprint, a score recommended by the European Commission that evaluates the environmental impact of a food product based on 16 indicators calculated throughout the life cycle of the products (e.g., climate change in kg carbon dioxide eq, marine eutrophication in kg N eq, land and water use or acidification in mol H+ eq).
  Instructions will introduce and explain the environmental label to the participants as "In the virtual supermarket, each product will have an environmental label. This label describes whether a product had a negative impact on the environment (green house gaz emissions, water resources depletion, etc.) from A, lowest impact, to E, highest impact.
  Arms: Environmental labelling

SUMMARY:
A 2-arm randomised control trial (with and without labels) will be conducted to test the effects of an environmental label on food choices in a virtual supermarket. A sample of 130 participants will take part in two shopping tasks: 1/ selection of 3 products to prepare a home-made dish, and 2/ selection of a ready-to-eat dish. These two tasks will be repeated for two scenarios: 1/ participants will be asked to select the foods for usual meals, and 2/ participants will be asked to select the foods for environmentally-friendly meals. This experimental design will allow to compare food choices in the presence vs. the absence of an environmental label and to investigate whether the label is informative and likely to help individuals to choose more environmental-friendly food options when explicitly asked to do so.

DETAILED DESCRIPTION:
See attached protocol documents

ELIGIBILITY:
Inclusion Criteria:

* Responsible for a substantial proportion of household grocery shopping
* Fluent in French

Exclusion Criteria:

* Dietary restrictions (vegetarian, vegan, allergies, intolerance, …)
* Uncorrected eye problems
* Known symptoms of nausea and dizziness when wearing a virtual reality headset

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Environmental impact of the food items selected | 15 minutes (the time frame denotes time taken to make the food choice task and there is no follow up)
  The environmental impact of the food selection will be calculated using the Product Environmental Footprint score for 100g of products throughout their life cycle.

SECONDARY OUTCOMES:
Familiarity for the food items selected | 15 minutes (the time frame denotes time taken to make the food choice task and there is no follow up)
  The familiarity for each food selected will be assessed using a discrete scale from 1 (never purchased) to 5 (very often purchased).
Liking for the food items selected | 15 minutes (the time frame denotes time taken to make the food choice task and there is no follow up)
  The liking for each food selected will be assessed using a discrete scale from 1 (I don't like it at all) to 10 (I like it very much).
Nutritional quality of the food items selected | 15 minutes (the time frame denotes time taken to make the food choice task and there is no follow up)
  The nutritional quality of the food selection will be calculated using the score from the British Food Standards Agency nutrient profiling system (FSA score).
Level of processing of the food items selected | 15 minutes (the time frame denotes time taken to make the food choice task and there is no follow up)
  The level of processing of the food selection will be estimated using a food classification system based on food processing (NOVA).
Price of the food items selected | 15 minutes (the time frame denotes time taken to make the food choice task and there is no follow up)
  Price of the food selection will be calculated per 100 kcal.

CONTACTS AND LOCATIONS:
Overall Officials: Lucile Marty, PhD, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre des Sciences du Goût et de l'Alimentation, Dijon, France

IPD SHARING:
Plan to Share IPD: Yes
Share on Open Science Framework
Supporting Information: Study Protocol, SAP
Time Frame: On publication, indefinitely
Access Criteria: Open website
URL: https://osf.io/du58k/

REFERENCES:
- [Derived] Arrazat L, Chambaron S, Arvisenet G, Goisbault I, Charrier JC, Nicklaus S, Marty L. Traffic-light front-of-pack environmental labelling across food categories triggers more environmentally friendly food choices: a randomised controlled trial in virtual reality supermarket. Int J Behav Nutr Phys Act. 2023 Jan 26;20(1):7. doi: 10.1186/s12966-023-01410-8. PMID 36703160
- Available data/document: Study Protocol — https://osf.io/du58k/
- Available data/document: Statistical Analysis Plan — https://osf.io/du58k/
- Available data/document: Individual Participant Data Set — https://osf.io/du58k/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT04909372/Prot_SAP_000.pdf